CLINICAL TRIAL: NCT02754154
Title: Real-World Comparative Observational Study in Non-Valvular Atrial Fibrillation Patients Using Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-433
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; apixaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients using Warfarin: Patients 18 years of age and older with Non-Valvular Atrial Fibrillation (NVAF) using Warfarin
  Interventions: Drug: Warfarin
- Patients using Apixaban: Patients 18 years of age and older with Non-Valvular Atrial Fibrillation (NVAF) using Apixaban
  Interventions: Drug: Apixaban
- Patients using Dabigatran: Patients 18 years of age and older with Non-Valvular Atrial Fibrillation (NVAF) using Dabigatran
  Interventions: Drug: Dabigatran
- Patients using Rivaroxaban: Patients 18 years of age and older with Non-Valvular Atrial Fibrillation (NVAF) using Rivaroxaban
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Warfarin
  Groups: Patients using Warfarin
Drug: Apixaban
  Groups: Patients using Apixaban
Drug: Dabigatran
  Groups: Patients using Dabigatran
Drug: Rivaroxaban
  Groups: Patients using Rivaroxaban

SUMMARY:
The purpose of this study is to compare the risk of major bleeding event among nonvalvular atrial fibrillation patients treated with warfarin, apixaban, dabigatran and rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old as of the index date
* At least 1 diagnosis of atrial fibrillation in the 12 months prior to or on index date, identified by any medical claim
* At least one year of baseline period and continuous enrollment for at least 12 months prior to index date Individuals with NVAF who were using oral anticoagulants (i.e., warfarin, dabigatran, rivaroxaban and apixaban) within the study period beginning Jan 1, 2012 through December 31, 2013 or last date of the last data cut available at the time of execution of the study

Exclusion Criteria:

* Patients with evidence of valvular heart disease, thyrotoxicosis, pericarditis, mitral stenosis, Venous thromboembolism(VTE), heart surgery, and endocarditis during the baseline period any time prior to or on index date
* Patients with any evidence of pregnancy at any time during the baseline will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older with Non-Valvular Atrial Fibrillation (NVAF) using oral anticoagulants
Sampling Method: Non-Probability Sample
Enrollment: 321182 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Time to "First Major" Bleeding event | Up to 25 months

SECONDARY OUTCOMES:
Time to "First Any" Bleeding event | Up to 25 months
Major Bleeding-Related Healthcare Utilization | Up to 25 months
  (Number of Hospitalizations, Total Length of Hospital Stay (days), Time to Hospitalization, Number Of Emergency Room (ER) visits, and Number of Outpatient Visits with at least 1 major bleeding event )
Any Bleeding-Related Healthcare Utilization | Up to 25 months
  (Number of Hospitalizations, Total Length of Hospital Stay (days), Time to Hospitalization, Number Of Emergency Room (ER) visits, and Number of Outpatient Visits with at least 1 bleeding event )
Major Bleeding-Related direct medical cost | Up to 25 months
  (Inpatient costs, Outpatient costs, and Emergency Room (ER) costs related to at least 1 major bleeding event)
Any Bleeding-Related direct medical cost | Up to 25 months
  (Inpatient costs, Outpatient costs, and Emergency Room (ER) costs related to at least 1 bleeding event)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm